CLINICAL TRIAL: NCT00921154
Title: A Single-dose, Randomised, Crossover Study to Compare the Rate and Extent of Absorption of Two Formulations of Ivermectin in Healthy, Fasting Male and Female Volunteers
Brief Title: Ivermectin Solution Bioequivalence Study - Fasted
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: SCO2704
Record Dates: First submitted 2009-06-15; First posted 2009-06-16 (Estimated); Last update posted 2011-10-06 (Estimated); Status verified 2011-10

CONDITIONS: Healthy
Keywords: therapeutic equivalency; pharmacokinetics; fasting; Healthy Volunteers
MeSH Terms: conditions — Fasting | interventions — Ivermectin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ivermectin (Experimental): Ivermectin
  Interventions: Drug: ivermectin

INTERVENTIONS:
Drug: ivermectin — Each subject will receive single doses of (i) 30 ml ivermectin oral solution (30 mg) and (ii) 10 x 3 mg tablets of ivermectin (30 mg) in 2 separate dosing periods with a 14 day wash-out period. Doses will be administered after an overnight fast.
  Other Names: Stromectol

SUMMARY:
The purpose of this study was to compare the pharmacokinetic and bioavailability profile (rate and amount of absorption into the bloodstream) of a test formulation of ivermectin solution 1 mg/ml with a marketed reference formulation of ivermectin 3 mg tablets when taken after an overnight fast .The study is designed in accordance with the EU Note for Guidance on the Investigation of Bioavailability and Bioequivalence 2001.

DETAILED DESCRIPTION:
Ivermectin is an antiparasitic medicine (i.e. a medicine used to eliminate parasitic worms) for oral administration, and is approved in the US and some other countries in a tablet form. A new liquid formulation of ivermectin has been developed to facilitate dosing. This is a single dose, randomised, crossover study in healthy adult male and female volunteers, with doses taken after an overnight fast. Doses will be separated by washout period of at least 14 days. Twenty-one blood samples will be taken from each volunteer over 144 hours in each period. Concentrations of ivermectin in plasma will be measured using a validated chromatographic assay (LC-MS/MS). Standard pharmacokinetic parameters will be obtained and bioequivalence on the basis of rate and extent of drug absorption will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* BMI <= 30 kg/m2 Weight between 50 and 90 kg
* Non-smokers, or smokers of fewer than 10 cigarettes per day
* Clinically normal medical history and physical exam findings
* Negative screening results for protocol-specified drugs of abuse
* Negative HIV and Hepatitis B and C tests
* Appropriate use of contraception and negative pregnancy test
* Ability to comprehend and communicate effectively with investigative staff
* Ability to give written informed consent

Exclusion Criteria:

* pregnant or nursing subjects
* subjects who lived in region endemic for certain parasitic worm diseases
* any protocol-specified vital sign or medical history that would preclude participation in the trial, including, but not limited to recent blood donation (or loss) and positive screens for HIV, Hepatitis B, or Hepatitis C
* Any indication of current or previous abuse of alcohol, solvents or drugs
* Intake of grapefruit products within 7 days before the start of the study
* Intake of methylxanthine-containing beverages within 24 hours prior to each study period or quantities of methylxanthine or alcohol-containing beverages which, in the opinion of the Investigator are abnormal (more than 5 cups or glasses of tea, coffee, cola, chocolate etc. per day or more than 20 g alcohol/day)
* Patients with a known or suspected intestinal helminth infection
* Patients with a known hypersensitivity to any component of the Ivermectin product.
* Smoking or alcohol consumption greater than protocol-specified levels
* Protocol-specified contraindication to blood sampling
* Acute or chronic medical, dietary or psychiatric condition or laboratory abnormality that may increase the risk associated with trial participation or investigational product administration or may interfere with the interpretation of trial results and, in the judgment of the investigator, would make the subject inappropriate for entry into this trial

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2005-03; Primary Completion 2005-05 (Actual); Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameters, including AUC0-t, AUC0-inf and Cmax | 21 samples over 144 hours in each period

SECONDARY OUTCOMES:
Pharmacokinetic parameters, including t1/2, Mean residence time, Terminal Elimination Rate Constant, and Tmax | 21 samples over 144 hours in each period

CONTACTS AND LOCATIONS:
Overall Officials: Jerry Cottrell, Study Director — McNeil UK
Locations (1):
- Shandon Clinic, Cork, Co. Cork, Ireland